CLINICAL TRIAL: NCT03274778
Title: An Exploratory proof-of Mechanism Study to Assess the Effect of Ruxolitinib on Tumor Infiltrating Myeloid Cells and Additional Immune Subsets in Prostate Cancer Patients
Brief Title: Effect of Ruxolitinib on Tumor Infiltrating Myeloid Cells
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty due to eligibility criteria.
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOSI-IOR-001
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Oral administration of Ruxolitinib 20mg BID for 28 consecutive days
  Interventions: Drug: Ruxolitinib 20 MG

INTERVENTIONS:
Drug: Ruxolitinib 20 MG — tablets
  Other Names: Jakavi

SUMMARY:
Ruxolitinib will be dispensed to patients candidate to prostatectomy immediately after histological diagnosis of prostate adenocarcinoma. The treatment will be given for 28 days followed by a prostatectomy thereafter.

Tumor material and blood samples will be analysed before, during and after the treatment with Ruxolitinib.

DETAILED DESCRIPTION:
Patients with suspected localized prostate cancer will undergo biopsies spotting different prostate sites, as per standard clinical practice. Patients with histologically confirmed prostate adenocarcinoma and candidate for prostatectomy, after signing the Informed Consent Form, will receive Ruxolitinib for 4 weeks (the time normally elapsing between histological diagnosis and surgery) and will thereafter undergo prostatectomy.

Remaining biological material from the diagnosis and the prostatectomy will be sent to the Molecular Oncology Laboratory for molecular analysis.

In addition, blood samples will be drawn before, during Ruxolitinib treatment (Week 2), at the end of treatment (Week 4), and after prostatectomy (Week 5), to assess the frequency and subtype of immune subsets and the circulating levels of cytokines and secreted.

Patients will be monitored for occurrence of adverse events/surgical complications during treatment and up to 4 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Histological diagnosis of prostate adenocarcinoma
* Stage ≥T2b for which surgery is indicated
* No distant metastasis (M0)
* NLR ≥3 in the blood or NLR ≥3 in the tumor biopsies or a percentage of MDSCs ≥ 30% in the tumour biopsies
* PS (ECOG scale) 0-1
* Adequate hepatic function: ALT and ASAT ≤ 2.5 x ULN, Bilirubin ≤ 1.5 ULN (exception if Gilbert's syndrome ≤ 2.5 x ULN)
* Adequate renal function: calculated creatinine clearance ≥ 50 ml/min according to the formula of Cockcroft-Gault
* Hemoglobin ≥ 10 g/dl, leukocyte count ≥ 4.0 x 103/µl, platelet count ≥ 200 x 103/µl
* Informed Consent as documented by the patient's signature

Exclusion Criteria:

* No history of coagulation disorders and normal INR
* Significant cardiovascular disorders in the last 12 months
* Other clinically significant concomitant disease states which in the opinion of the Investigator may represent contraindications to study participation
* Known or suspected non-compliance
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Ongoing treatment with strong CYP3A4 inhibitors or dual CYP2C9 and CYP3A4 inhibitors

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Tumor immune response | 9 wks
  Tumor immune response modification induced by Ruxolitinib

SECONDARY OUTCOMES:
pSTAT3 | 5 wks
  Decrease of pSTAT3
Cytokines | 6 wks
  Reduction of cytokines associated to myeloid cells recruitment and tumor-promoting factors (e.g. IL8, IL6, TGF)
KI-67 | 9 wks
  Reduction by 50% of KI-67
biomarkers | 5 wks
  Increase of senescence and apoptosis markers (p16, p21, Beta-galactosidase, Caspase-3, Caspase-8)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Alimonti, Prof., Study Director — Institute of Oncology Research (IOR)
Locations (1):
- Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No